CLINICAL TRIAL: NCT00703144
Title: Pharmacokinetics of Piperacillin and Tazobactam in Anuric Septic Patients Treated by Continuous Veno Venous Hemodiafiltration
Brief Title: Pharmacokinetics of Piperacillin/Tazobactam in Patients Treated by Continuous Renal Replacement Therapy
Acronym: PTCRRT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07 300 02; University Hospital Toulouse
Record Dates: First submitted 2008-06-20; First posted 2008-06-23 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Diffusive and Convective Clearance; Body Clearance; Piperacillin Tazocilline Concentrations (Cmin)
Keywords: Pharmacokinetics; piperacillin/tazobactam.; Septic patients; oliguric renal failure; continuous veno-venous hemodiafiltration.
MeSH Terms: interventions — Piperacillin, Tazobactam Drug Combination; Pharmacogenomic Variants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pharmacokinetic (Experimental)
  Interventions: Drug: piperacillin/tazobactam; Procedure: Pharmacokinetic

INTERVENTIONS:
Drug: piperacillin/tazobactam — piperacillin 4 g and tazobactam 500 mg during 30 min IV infusion every 8h during 2 consecutive days
  Other Names: Tazocilline
Procedure: Pharmacokinetic

SUMMARY:
The pharmacokinetics of piperacillin/tazobactam will be evaluated in twenty septic patients with renal failure undergoing continuous veno-venous hemodiafiltration.

DETAILED DESCRIPTION:
The pharmacokinetics of piperacillin/tazobactam will be evaluated in twenty septic patients with renal failure undergoing continuous veno-venous hemodiafiltration. This is a prospective study.

Continuous replacement therapy has a continuous effect on drug elimination which could compromise effective antibiotic treatment.

Patients will receive a standard course of pip/tazo 4g intravenously 8 hourly administrated immediately when CVVHDF will be started.

Blood samples will be collected at 30mn, 2h, 4h, 6h, 8h, 16h, 24h for the first and the second day.

We will measure plasma piperacillin/tazobactam concentration and compare them to MICs for the whole dosing interval.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older .
* Females of childbearing potential must have a negative pregnancy test at screening.
* Subjects whose life expectancy is estimated over 7 days.
* Anuric patients requiring continuous venovenous hemodiafiltration
* Septic patients,severe sepsis or septic shock
* Written informed consent should be given either by the patient or a member of his family

Exclusion Criteria:

* Subjects with a history of true allergy or adverse drug reactions
* Pathogens whose antibiotic susceptibility is not proved.
* Patients having impaired hepatic function
* Contraindication of anticoagulation by heparin
* Residual renal function
* Participation in a clinical trial
* Interruption of treatment by piper/tazo or hemodiafiltration during the study.
* Patients with psychiatric disorder or serious medical condition which in the opinion of the investigator may lead to complexity in patient management.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Serum levels of both piperacillin and tazobactam (Cmin) during 2 daus | 2 days

SECONDARY OUTCOMES:
Body clearance | 2 days

CONTACTS AND LOCATIONS:
Overall Officials: LAVAYSSIERE Laurence, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Service de Néphrologie, Toulouse, France